CLINICAL TRIAL: NCT02535858
Title: Virtual Environment With Biofeedback to Promote Awareness of Relapse Risk Among Chemically Dependent Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Annie France Frère Slaets, PhD, University of Mogi das Cruzes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0094.0.237.000-07
Record Dates: First submitted 2015-08-10; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Anxiety
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Respiratory Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart and respiratory rate and video (Experimental): To determine the limits between normal and emotional anxious, thirty volunteers male's adults (GL) with age range between 20 and 50 years were recruited. None of them had any pathology associated with anxiety or psychiatric disorders, and none was drugs user or taking medication.
  Interventions: Device: Heart and respiratory rate and video
- Heart and respiratory rate and VE (Experimental): A second group has fifty adult volunteers (DG) ongoing outpatient chemical dependency clinic [treatment average's population: 5 months and 14 days]. The patients were abstained from drugs use for at least two months, and they were selected to test the VE. None of the DG's participants had any pathology associated with anxiety or psychiatric disorders, and none was taking medications. The DG volunteers were narcotic users of two or more illicit drugs, such as alcohol, marijuana, tobacco, cocaine and crack cocaine. Addiction for alcohol and tobacco were 72% and 56% respectively. The group's percentage for using psychoactive drugs were, 70% for cocaine and crack cocaine and 32% for marijuana.
  Interventions: Device: Heart and respiratory rate and VE

INTERVENTIONS:
Device: Heart and respiratory rate and VE — To evaluate the effectiveness of the virtual environment (VE) as a biofeedback of chemically dependent's vulnerability front situations of risk, a total of 50 volunteers who were drug users, monitored by 10 therapists, were enrolled.
  Arms: Heart and respiratory rate and VE
Device: Heart and respiratory rate and video — Anxiety is characterized by the average variability from both heart and respiratory rate of 30 volunteers undergoing stress environment situations.
  Arms: Heart and respiratory rate and video

SUMMARY:
Anxiety is one of the major influences on relapse and substance abuse treatment dropout. Chemically dependent individuals need to be aware of their emotional state in situations that jeopardise their treatment. The current therapeutic resources still subjective and with limited treatment success. This research presents a developed virtual environment (VE) simultaneously connected to a physiological signals device acquisition that allows, through a biofeedback, the chemically dependents consciousness on their vulnerability front different situations of 'risk', without a direct assessment of the therapist. Developed in 3ds Max® software, the VE is composed of scenarios and objects that are in the habit of the chemically dependent individual's daily life. The interaction with the environment is accomplished using a Human-Computer Interface (HCI) that converts incoming physiological signals indicating anxiety state into commands that change the scenes. Anxiety is characterized by the average variability from both heart and respiratory rate of 30 volunteers undergoing stress environment situations. To evaluate the effectiveness of the VE as a biofeedback of chemically dependent's vulnerability front situations of risk, a total of 50 volunteers who were drug users, monitored by 10 therapists, were enrolled. Prior VE, the results demonstrated a poor correlation between the therapists' predictions and those of the chemically dependent individuals. After exposure to the VE, there was a significant increase of 73% in awareness of the risks of relapse by the chemically dependent individuals, confirming the hypothesis that the VE coupled to the biofeedback device may assist the therapist with treatment.

DETAILED DESCRIPTION:
2.1 Ethical approval Approval was obtained from the Local Ethics Committee (CAAE-0094.0.237.000-07, process CEP/UMC-093/2007) for the participants. They had been informed about the methodology and confidentiality of their personal information. The participants were informed about the methodology and confidentiality of their personal information. All procedures were performed after written informed consent from all participants.

2.2 Study Participants To determine the limits between normal and emotional anxious, thirty volunteers male's adults (GL) with age range between 20 and 50 years were recruited. None of them had any pathology associated with anxiety or psychiatric disorders, and none was drugs user or taking medication. Three mental health professionals (PG1), specialized in chemical dependency, evaluated the emotional state of the volunteers.

A second group has fifty adult volunteers (DG) (mean age of 35±10.02 years) ongoing outpatient chemical dependency clinic [treatment average's population: 5 months and 14 days]. The patients were abstained from drugs use for at least two months, and they were selected to test the VE. None of the DG's participants had any pathology associated with anxiety or psychiatric disorders, and none was taking medications. The DG volunteers were narcotic users of two or more illicit drugs, such as alcohol, marijuana, tobacco, cocaine and crack cocaine. Addiction for alcohol and tobacco were 72% and 56% respectively. The group's percentage for using psychoactive drugs were, 70% for cocaine and crack cocaine and 32% for marijuana.

For this group, 10 mental health professionals (PG2), therapists, specialized in chemical dependency and responsible for monitoring the group's treatment assessed their emotional states.

To elaborate the scenarios and characterize the characters in the virtual environment (VE), another eight specialists professionals (PG3) from the chemical dependency field recommended situations, places, objects, signs, or cues thought to trigger craving.

2.4 Testing Protocol Prior CDI to the test, the therapist answered a questionnaire identifying the situations of risk presented in the VE that could lead the patient to relapse. The same questionnaire was also completed by the CDI before and after the VE test. In addition, this application was structured based on risk factors survey.

The questions presented are listed below:

1. If you receive a phone call from a friend that is a drug user, would it stimulate you to take drugs?
2. If you walk on places that used to be selling drugs areas, would you relapse by any chance?
3. If a colleague invites you to have drinks, would you be favored by taking drugs?
4. Family issues or situations where the family is absent, would it contribute to your relapse?
5. Would you relapse if you had the chance of going party or places that might have drugs?
6. A friendship that is a drug user and can offer it to you would trigger your wishes for having drugs? The questionnaire and VE test were applied to each CDI in a single day on mornings. The patients were present with their therapists while performing the test.

The test was conducted in a comfortable room that was part of a therapeutic community for CDIs. This room held the test equipment, a support table for the equipment, and chairs for the patient and therapist. Communication during the test was not recommended. Extra care was taken to avoid tests' interruptions including disturbance caused by equipment (air conditioning, audio, etc.) as well as people entering at the exam room. Regarding the sensors, the cardiac frequency meter was placed on the distal phalanx of the little finger and the respiratory rate (RR) sensor near the right nostril using a headset support. The CDIs were informed that the outcome of each situation presented in the VE would correspond to their physiological state when facing the risk situations. Their questions were answered, and only their emotions were shown to influence the scenarios. The test started with the volunteers watching a desired film selected by themselves where the basal levels from both physiological signals were simultaneously acquired. It was followed by the introduction of the developed VE where both heart and respiratory rates were measured between minutes and compared with the previously acquired baseline levels. The script automatically selected the scenes depending on the identified emotional state. When the state was identified as anxious, the program changed the scene, showing the character using drugs. Otherwise, the plot proceeded.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers (DG) ongoing outpatient chemical dependency clinic [treatment average's population: 5 months and 14 days].
* The patients were abstained from drugs use for at least two months, and they were selected to test the VE.
* None of the DG's participants had any pathology associated with anxiety or psychiatric disorders, and none was taking medications.
* The DG volunteers were narcotic users of two or more illicit drugs, such as alcohol, marijuana, tobacco, cocaine and crack cocaine.

Exclusion Criteria:

* The patients were not abstained from drugs use for at least two months

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Percentage of the variation in respiratory and heart rate. | The respiratory and heart rate were collected during 10 minutes from each no-drugs user and 30 minutes from each chemically dependent individual.
  This research presents a developed virtual environment (VE) simultaneously connected to a physiological signals device acquisition (heart and respiratory rates) that allows, through a biofeedback, the chemically dependents consciousness on their vulnerability front different situations of 'risk', without a direct assessment of the therapist. During the virtual exposure, the heart and respiratory rates of the chemically dependent individual (CDI) were acquired and processed to be classified as a normal or anxious state. Then, the scenes were automatically changed depending on the captured physiological signals. The signals' average were calculated for each individual and emotional state (normal vs. anxious). A volunteer was considered to be anxious if the heart or respiratory rates are at least 7% and 16% above the basal levels respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Annie F. Frère, PhD, Principal Investigator — University of Mogi Cruzes
Locations (1):
- University of Mogi das Cruzes, Mogi das Cruzes, São Paulo, Brazil